CLINICAL TRIAL: NCT01668017
Title: A Multicentre, Open Label, Phase I Trial in Japan of the MEK Inhibitor Pimasertib Given Orally to Subjects With Solid Tumors as Monotherapy
Brief Title: A Multicentre, Open Label, Phase 1 Trial in Japan of the Mitogen Activated Protein Extracellular Signal Regulated Kinase (MEK) Inhibitor Pimasertib Given Orally to Subjects With Solid Tumors as Monotherapy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The sponsor decided not to conduct the expansion part of trial (part 2)
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono Co., Ltd., Japan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR 200066-010
Record Dates: First submitted 2012-08-15; First posted 2012-08-17 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2017-08-23 (Actual); Status verified 2017-07

CONDITIONS: Advanced Solid Tumors; Hepatocellular Carcinoma
Keywords: Advanced solid tumors; Hepatocellular carcinoma; cancer, liver
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — N-(2,3-dihydroxypropyl)-1-((2-fluoro-4-iodophenyl)amino)isonicotinamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Part 1: Pimasertib 30mg in Solid Tumor (Experimental)
  Interventions: Drug: Pimasertib
- Part 1: Pimasertib 45 mg in Solid Tumor (Experimental)
  Interventions: Drug: Pimasertib
- Part 1: Pimasertib 60 mg in Solid Tumor (Experimental)
  Interventions: Drug: Pimasertib
- Part 1: Pimasertib 30 mg in Hepatocellular Carcinoma (HCC) (Experimental)
  Interventions: Drug: Pimasertib
- Part 1: Pimasertib 45 mg in HCC (Experimental)
  Interventions: Drug: Pimasertib

INTERVENTIONS:
Drug: Pimasertib — Subjects with solid tumor will be administered with Pimasertib 30 mg twice a day (BID) in 21-day cycles until disease progression, intolerable toxicity, investigators decision to discontinue treatment or withdrawal of consent by the subject.
  Arms: Part 1: Pimasertib 30mg in Solid Tumor
Drug: Pimasertib — Subjects with solid tumor will be administered with Pimasertib 45 mg BID in 21-day cycles until disease progression, intolerable toxicity, investigators decision to discontinue treatment or withdrawal of consent by the subject.
  Arms: Part 1: Pimasertib 45 mg in Solid Tumor
Drug: Pimasertib — Subjects with solid tumor will be administered with Pimasertib 60 mg BID in 21-day cycles until disease progression, intolerable toxicity, investigators decision to discontinue treatment or withdrawal of consent by the subject.
  Arms: Part 1: Pimasertib 60 mg in Solid Tumor
Drug: Pimasertib — Subjects with HCC will be administered with Pimasertib 30 mg BID in 21-day cycles until disease progression, intolerable toxicity, investigators decision to discontinue treatment or withdrawal of consent by the subject.
  Arms: Part 1: Pimasertib 30 mg in Hepatocellular Carcinoma (HCC)
Drug: Pimasertib — Subjects with HCC will be administered with Pimasertib 45 mg BID in 21-day cycles until disease progression, intolerable toxicity, investigators decision to discontinue treatment or withdrawal of consent by the subject.
  Arms: Part 1: Pimasertib 45 mg in HCC

SUMMARY:
This is a two-part trial. "Solid tumor" in this protocol means solid tumor excluding hepatocellular carcinoma (HCC).

Part 1: Dose Escalation Phase in subjects with solid tumor (Cohort A) and HCC (Cohort B). The dose will be increased from 45 mg twice a day (BID) with 3+3 cohort method up to the recommended phase 2 dose (RP2D) of pimasertib established as single agent in the global studies for each arm independently.

Part 2: The Maximum Tolerated Dose (MTD) defined in Part 1 will be confirmed in more subjects in Cohort A (N=18) and Cohort B (N=6) separately.

Following the recommendation by the Safety Monitoring Committee, Cohort B was discontinued due to hepatocellular carcinoma (HCC) and there will be no further enrollment of subjects to this cohort. This decision is based upon review of safety and efficacy information.

ELIGIBILITY:
Inclusion Criteria:

Cohort A: A histologically or cytologically confirmed diagnosis of advanced solid tumors which is either refractory after standard therapy for the disease or for which no effective standard therapy is available. Archived tumor tissue available or biopsy of tumor tissue needs to be performed.

Cohort B: A histologically or cytologically confirmed diagnosis of advanced hepatocellular carcinoma (HCC) which is either refractory after standard therapy for the disease or for which no effective standard therapy is available. Archived tumor tissue available or biopsy of tumor tissue needs to be performed. Subjects with Child Pugh A.

* Male or female Japanese, age greater than or equal to (>=) 18 years.
* Subject has read and understands the informed consent form and is willing and able to give informed consent. The subject fully understands requirements of the trial and is willing to comply with all trial visits and assessments.
* Women of childbearing potential must have a negative blood pregnancy test at the screening visit.
* Female subjects of childbearing potential and male subjects with female partners of childbearing potential must be willing to avoid pregnancy by using an adequate method of contraception for 2 weeks prior to, during and four weeks after the last dose investigational medicinal product (IMP).
* Life expectancy of at least 3 months

Exclusion Criteria:

Hematological abnormality Cohort A: Hematological test abnormalities of Hemoglobin < 9.0 g/dL, Neutrophil count < 1.0*10^9/L and Platelet count < 100*10^9/L.

Cohort B: Hematological test abnormalities of Hemoglobin < 9.0 g/dL, Neutrophil count < 1.0*10^9/L, Platelet count < 75*10^9/L, subjects with hepatic encephalopathy

* Renal impairment as evidenced by serum creatinine > 1.5*upper limit of normal (ULN), and calculated creatinine clearance < 60 mL/min by Cockcroft-Gault formula.
* Liver function abnormality of Total Bilirubin > 1.5*ULN, or aspartate transaminase 9AST) or alkaline phosphatase (ALT)> 2.5*ULN. For subjects with HCC or liver involvement AST/ALT > 5*ULN.
* History of central nervous system (CNS) metastases, unless subject has been previously treated for CNS metastases
* History of difficulty swallowing, malabsorption or other chronic gastro-intestinal disease or conditions
* Eastern Cooperative Oncology Group Performance status (ECOG PS) greater than 1.
* Has received chemotherapy, immunotherapy, hormonal therapy, biologic therapy, or any other anticancer therapy (including any investigational agent) or surgical intervention within 28 days or 5 half lives for non-cytotoxics of registration.
* Baseline corrected QT interval on screening ECG (QTc) >= 480 ms or left ventricular ejection fraction (LVEF) < 40% on screening echocardiogram
* Cohort B: Subjects with hepatic encephalopathy, remarkable ascites and subjects with history of esophageal varices rupture within 6 months (subjects with symptom improvement after treatment are eligible)
* Other serious illness or medical conditions.
* Retinal degenerative disease.
* Previous treatment with MEK inhibitors.
* Legal incapacity or limited legal capacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-09-30 (Actual); Primary Completion 2015-05-31 (Actual); Study Completion 2015-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Serono Co., Ltd., Tokyo, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- Please contact, Merck Serono Co., Ltd For Recruiting Locations in, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First/last subject (informed consent): September 2012/April 2015. Last subject completed: April 2015.
Pre-assignment Details: This study was to be conducted in 2 parts; Part 1 was the dose escalation phase and Part 2 was the expansion phase. However, due to early termination of the study, the sponsor decided not to conduct the expansion phase (Part 2).
Groups:
- Part 1: Pimasertib 30 mg in Solid Tumor: Subjects with solid tumor were administered with Pimasertib 30 milligram (mg) twice a day (BID) in 21-day cycles until disease progression, intolerable toxicity, investigators decision to discontinue treatment or withdrawal of consent by the subject.
- Part 1: Pimasertib 45 mg in Solid Tumor: Subjects with solid tumor were administered with Pimasertib 45 mg BID in 21-day cycles until disease progression, intolerable toxicity, investigators decision to discontinue treatment or withdrawal of consent by the subject.
- Part 1: Pimasertib 60 mg in Solid Tumor: Subjects with solid tumor were administered with Pimasertib 60 mg BID in 21-day cycles until disease progression, intolerable toxicity, investigators decision to discontinue treatment or withdrawal of consent by the subject.
- Part 1: Pimasertib 30 mg in Hepatocellular Carcinoma (HCC): Subjects with HCC were administered with Pimasertib 30 mg BID in 21-day cycles until disease progression, intolerable toxicity, investigators decision to discontinue treatment or withdrawal of consent by the subject.
- Part 1: Pimasertib 45 mg in HCC: Subjects with HCC were administered with Pimasertib 45 mg BID in 21-day cycles until disease progression, intolerable toxicity, investigators decision to discontinue treatment or withdrawal of consent by the subject.
Period: Overall Study
Arm/Group | Part 1: Pimasertib 30 mg in Solid Tumor | Part 1: Pimasertib 45 mg in Solid Tumor | Part 1: Pimasertib 60 mg in Solid Tumor | Part 1: Pimasertib 30 mg in Hepatocellular Carcinoma (HCC) | Part 1: Pimasertib 45 mg in HCC
Started | 4 | 9 | 6 | 5 | 2
Completed | 4 | 9 | 6 | 5 | 2
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all subjects who received at least one administration of pimasertib.
Groups:
- Part 1: Pimasertib 30 mg in Solid Tumor: Subjects with solid tumor were administered with Pimasertib 30 mg BID in 21- day cycles until disease progression, intolerable toxicity, investigators decision to discontinue treatment or withdrawal of consent by the subject.
- Part 1: Pimasertib 30 mg in HCC: Subjects with HCC were administered with Pimasertib 30 mg BID in 21-day cycles until disease progression, intolerable toxicity, investigators decision to discontinue treatment or withdrawal of consent by the subject.
- Total: Total of all reporting groups
Arm/Group | Part 1: Pimasertib 30 mg in Solid Tumor | Part 1: Pimasertib 45 mg in Solid Tumor | Part 1: Pimasertib 60 mg in Solid Tumor | Part 1: Pimasertib 30 mg in HCC | Part 1: Pimasertib 45 mg in HCC | Total
Number analyzed (Participants) | 4 | 9 | 6 | 5 | 2 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (12.20) | 61.4 (10.63) | 61.5 (9.29) | 58.8 (13.63) | 56.5 (20.51) | 60.7 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 4 | 2 | 1 | 13
  Male | 2 | 5 | 2 | 3 | 1 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Experienced at Least One Dose Limiting Toxicity (DLT)
Description: DLT defined using National Cancer Institute Common Toxicity Criteria for Adverse Events Version 3.0 (NCI CTCAE v3.0): any of following toxicities possibly/probably related to study drug: Any non-hematological toxicity of Grade 3 or higher (excluding Grade 3 asymptomatic rise in liver function tests (aspartate aminotransferase [AST], alanine aminotransferase [ALT], alkaline phosphatase [ALP], gamma-glutamyl transferase [GGT] reversible in 7 days for subjects with solid tumor and without liver involvement, or Grade 4 for subjects with HCC or with liver involvement; Grade 3 or 4 asymptomatic rise in creatinine phosphokinase (CPK) reversible in 7 days, deniable for myocardial infarction and rhabdomyolysis; Grade 3 vomiting/diarrhea encountered without optimal therapy). Any Grade 4 neutropenia >5 days duration, any Grade 3 or above febrile neutropenia. Grade 4 thrombocytopenia >1 day or Grade 3 with bleeding. Any treatment delay >2 weeks due to drug-related adverse effects.
Time Frame: During Treatment Cycle 1 (Day 1 to 21)
Population: DLT analysis set included all subjects who experienced any DLT during Cycle 1 and who received above 85% of all planned doses of pimasertib during Cycle 1.
Measure: Number; unit: subjects
Groups:
- Part 1: Pimasertib 30 mg in Solid Tumor: Subjects with solid tumor were administered with Pimasertib 30 mg BID in 21-day cycles until disease progression, intolerable toxicity, investigators decision to discontinue treatment or withdrawal of consent by the subject.
- Part 1: Pimasertib 60 mg in Solid Tumor: Subjects with solid tumor were administered with Pimasertib 60 mg BID in 21-day cycles until disease progression, intolerable toxicity, investigators decision to discontinue treatment or withdrawal of consent by the subject, whichever comes first.
- Part 1: Pimasertib 30 mg in HCC: Subjects with HCC were administered with Pimasertib 30 mg BID in 21-day cycles until disease progression, intolerable toxicity, investigators decision to discontinue treatment or withdrawal of consent by the subject, whichever comes first.
- Part 1: Pimasertib 45 mg in HCC: Subjects with HCC were administered with Pimasertib 45 mg BID in 21-day cycles until disease progression, intolerable toxicity, investigators decision to discontinue treatment or withdrawal of consent by the subject, whichever comes first.
Arm/Group | Part 1: Pimasertib 30 mg in Solid Tumor | Part 1: Pimasertib 45 mg in Solid Tumor | Part 1: Pimasertib 60 mg in Solid Tumor | Part 1: Pimasertib 30 mg in HCC | Part 1: Pimasertib 45 mg in HCC
Number analyzed (Participants) | 3 | 6 | 3 | 3 | 1
subjects | 0 | 0 | 2 | 1 | 1

2. Secondary Outcome: Number of Subjects Who Experienced Treatment-Emergent Adverse Events (TEAEs) or Serious TEAEs
Description: An adverse event (AE) was defined as any untoward medical occurrence which does not necessarily have a causal relationship with this the study drug. An AE was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug or worsening of pre-existing medical condition, whether or not related to study drug. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. Treatment-emergent are events between first dose of study drug and up to 30 days after last dose that were absent before treatment or that worsened relative to pre-treatment state. TEAEs include both Serious TEAEs and non-serious TEAEs.
Time Frame: Baseline up to 30 days post last dose of study drug; assessed maximum up to 39.4 weeks
Population: Safety analysis set included all subjects who received at least one administration of pimasertib.
Measure: Number; unit: subjects
Arm/Group | Part 1: Pimasertib 30 mg in Solid Tumor | Part 1: Pimasertib 45 mg in Solid Tumor | Part 1: Pimasertib 60 mg in Solid Tumor | Part 1: Pimasertib 30 mg in HCC | Part 1: Pimasertib 45 mg in HCC
Number analyzed (Participants) | 4 | 9 | 6 | 5 | 2
subjects
  TEAEs | 4 | 9 | 6 | 5 | 2
  Serious TEAEs | 2 | 2 | 2 | 2 | 0

3. Secondary Outcome: Maximum Observed Concentration (Cmax) of Pimasertib on Cycle 1 Day 1
Time Frame: Cycle 1: Pre-morning dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8, hours post dose, pre-evening dose (Hour 12) at Day 1
Population: Pharmacokinetic (PK) analysis set included all subjects who received at least 1 planned dose of pimasertib and who had at least 1 measurable post-dose concentration. Subjects with important protocol deviations or events, which may impact the quality of the PK data were excluded from the PK analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part 1: Pimasertib 30 mg in Solid Tumor | Part 1: Pimasertib 45 mg in Solid Tumor | Part 1: Pimasertib 60 mg in Solid Tumor | Part 1: Pimasertib 30 mg in HCC
Number analyzed (Participants) | 4 | 9 | 6 | 5
nanogram per milliliter (ng/mL) | 162.4 (113.1) | 222.1 (45.2) | 288.3 (52.1) | 167.6 (26.3)

4. Secondary Outcome: Maximum Observed Concentration (Cmax) of Part 1: Pimasertib 45 mg in HCC Arm on Cycle 1 Day 1
Description: The summarized data was not available for this arm therefore individual data was presented.
Time Frame: Cycle 1: Pre-morning dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8, hours post dose, pre-evening dose (Hour 12) at Day 1
Population: PK analysis set included all subjects who received at least 1 planned dose of pimasertib and who had at least 1 measurable post-dose concentration. Subjects with important protocol deviations or events, which may impact the quality of the PK data were excluded from the PK analysis set.
Measure: Number; unit: ng/mL
Arm/Group | Part 1: Pimasertib 45 mg in HCC
Number analyzed (Participants) | 2
ng/mL
  Subject 1 | 225
  Subject 2 | 281

5. Secondary Outcome: Maximum Observed Concentration (Cmax) of Pimasertib on Cycle 1 Day 15
Description: Data were not reported for "Part 1: Pimasertib 45 mg in HCC" arm as there were no PK samples collected for this arm.
Time Frame: Cycle 1: Pre-morning dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8, hours post dose, pre-evening dose (Hour 12) at Day 15
Population: PK analysis set. Here "Overall Number of Participants Analyzed" signifies the overall number of subjects who were evaluable for this outcome measure for each arm, respectively.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1: Pimasertib 30 mg in Solid Tumor | Part 1: Pimasertib 45 mg in Solid Tumor | Part 1: Pimasertib 60 mg in Solid Tumor | Part 1: Pimasertib 45 mg in HCC
Number analyzed (Participants) | 4 | 6 | 5 | 0
ng/mL | 199.5 (58.9) | 231.6 (66.1) | 336.3 (30.8) |

6. Secondary Outcome: Maximum Observed Concentration (Cmax) of Part 1: Pimasertib 30 mg in HCC Arm on Cycle 1 Day 15
Description: The summarized data was not available for this arm therefore individual data was presented.
Time Frame: Cycle 1: Pre-morning dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8, hours post dose, pre-evening dose (Hour 12) at Day 15
Population: as for outcome 4
Measure: Number; unit: ng/mL
Arm/Group | Part 1: Pimasertib 30 mg in HCC
Number analyzed (Participants) | 2
ng/mL
  Subject 1 | 320
  Subject 2 | 419

7. Secondary Outcome: Time to Reach Maximum Concentration (Tmax) on Cycle 1 Day 1
Time Frame: Cycle 1: Pre-morning dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8, hours post dose, pre-evening dose (Hour 12) at Day 1
Population: as for outcome 4
Measure: Median (Full Range); unit: hours
Arm/Group | Part 1: Pimasertib 30 mg in Solid Tumor | Part 1: Pimasertib 45 mg in Solid Tumor | Part 1: Pimasertib 60 mg in Solid Tumor | Part 1: Pimasertib 30 mg in HCC
Number analyzed (Participants) | 4 | 9 | 6 | 5
hours | 2.450 [0.48 to 4.00] | 1.480 [0.48 to 7.98] | 1.710 [0.97 to 2.43] | 1.000 [0.95 to 2.57]

8. Secondary Outcome: Time to Reach Maximum Concentration (Tmax) of Part 1: Pimasertib 45 mg in HCC Arm on Cycle 1 Day 1
Description: The summarized data was not available for this arm therefore individual data was presented.
Time Frame: Cycle 1: Pre-morning dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8, hours post dose, pre-evening dose (Hour 12) at Day 1
Population: as for outcome 4
Measure: Number; unit: hours
Arm/Group | Part 1: Pimasertib 45 mg in HCC
Number analyzed (Participants) | 2
hours
  Subject 1 | 1.47
  Subject 2 | 1.92

9. Secondary Outcome: Time to Reach Maximum Concentration (Tmax) on Cycle 1 Day 15
Description: Data were not reported for "Part 1: Pimasertib 45 mg In HCC" arm as there were no PK samples collected for this arm.
Time Frame: Cycle 1: Pre-morning dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8, hours post dose, pre-evening dose (Hour 12) at Day 15
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Arm/Group | Part 1: Pimasertib 30 mg in Solid Tumor | Part 1: Pimasertib 45 mg in Solid Tumor | Part 1: Pimasertib 60 mg in Solid Tumor | Part 1: Pimasertib 45 mg in HCC
Number analyzed (Participants) | 4 | 6 | 5 | 0
hours | 1.805 [1.00 to 2.48] | 1.910 [1.00 to 2.48] | 2.550 [1.50 to 5.88] |

10. Secondary Outcome: Time to Reach Maximum Concentration (Tmax) of Part 1: Pimasertib 30 mg in HCC Arm on Cycle 1 Day 15
Description: The summarized data was not available for this arm therefore individual data was presented.
Time Frame: Cycle 1: Pre-morning dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8, hours post dose, pre-evening dose (Hour 12) at Day 15
Population: as for outcome 4
Measure: Number; unit: hours
Arm/Group | Part 1: Pimasertib 30 mg in HCC
Number analyzed (Participants) | 2
hours
  Subject 1 | 0.98
  Subject 2 | 0.95

11. Secondary Outcome: Area Under the Concentration Over Time (AUCt) at Cycle 1 Day 1
Time Frame: Cycle 1: Pre-morning dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8, hours post dose, pre-evening dose (Hour 12) at Day 1
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 1: Pimasertib 30 mg in Solid Tumor | Part 1: Pimasertib 45 mg in Solid Tumor | Part 1: Pimasertib 60 mg in Solid Tumor | Part 1: Pimasertib 30 mg in HCC
Number analyzed (Participants) | 4 | 9 | 6 | 5
h*ng/mL | 703.0 (73.8) | 862.4 (42.8) | 1626.9 (43.6) | 911.4 (27.3)

12. Secondary Outcome: Area Under the Concentration Over Time (AUCt) of Part 1: Pimasertib 45 mg in HCC Arm on Cycle 1 Day 1
Description: The summarized data was not available for this arm therefore individual data was presented.
Time Frame: Cycle 1: Pre-morning dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8, hours post dose, pre-evening dose (Hour 12) at Day 1
Population: as for outcome 4
Measure: Number; unit: h*ng/mL
Arm/Group | Part 1: Pimasertib 45 mg in HCC
Number analyzed (Participants) | 2
h*ng/mL
  Subject 1 | 1754
  Subject 2 | 1430

13. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero up to Time Tau (AUC0-tau) of Pimasertib at Cycle 1 Day 1
Description: Area under the concentration-time curve from time zero up to time Tau, where Tau is the dosing interval (12 hours).
Time Frame: Cycle 1: Pre-morning dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8, hours post dose, pre-evening dose (Hour 12) at Day 1
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 1: Pimasertib 30 mg in Solid Tumor | Part 1: Pimasertib 45 mg in Solid Tumor | Part 1: Pimasertib 60 mg in Solid Tumor | Part 1: Pimasertib 30 mg in HCC
Number analyzed (Participants) | 3 | 8 | 6 | 5
h*ng/mL | 618.3 (86.1) | 857.4 (46.0) | 1629.3 (43.7) | 911.7 (27.2)

14. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero up to Time Tau (AUC0-tau) of Pimasertib of 1 Part 1: Pimasertib 45 mg in HCC Arm on Cycle 1 Day 1
Description: Area under the concentration-time curve from time zero up to time Tau, where Tau is the dosing interval (12 hours). The summarized data was not available for this arm therefore individual data was presented.
Time Frame: Cycle 1: Pre-morning dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8, hours post dose, pre-evening dose (Hour 12) at Day 1
Population: as for outcome 4
Measure: Number; unit: h*ng/mL
Arm/Group | Part 1: Pimasertib 45 mg in HCC
Number analyzed (Participants) | 2
h*ng/mL
  Subject 1 | 1761
  Subject 2 | 1431

15. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero up to Time Tau (AUC0-tau) of Pimasertib at Cycle 1 Day 15
Description: Area under the concentration-time curve from time zero up to time Tau, where Tau is the dosing interval (12 hours). Data were not reported for "Part 1: Pimasertib 45 mg In HCC" arm as there were no PK samples collected for this arm.
Time Frame: Cycle 1: Pre-morning dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8, hours post dose, pre-evening dose (Hour 12) at Day 15
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 1: Pimasertib 30 mg in Solid Tumor | Part 1: Pimasertib 45 mg in Solid Tumor | Part 1: Pimasertib 60 mg in Solid Tumor | Part 1: Pimasertib 45 mg in HCC
Number analyzed (Participants) | 4 | 6 | 4 | 0
h*ng/mL | 1189.3 (73.6) | 1125.0 (62.1) | 2140.7 (37.6) |

16. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero up to Time Tau (AUC0-tau) of Part 1: Pimasertib 30 mg in HCC Arm on Cycle 1 Day 15
Description: as for outcome 14
Time Frame: Cycle 1: Pre-morning dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8, hours post dose, pre-evening dose (Hour 12) at Day 15
Population: as for outcome 4
Measure: Number; unit: h*ng/mL
Arm/Group | Part 1: Pimasertib 30 mg in HCC
Number analyzed (Participants) | 2
h*ng/mL
  Subject 1 | 2250
  Subject 2 | 1687

17. Secondary Outcome: Apparent Terminal Half-life (t1/2) of Pimasertib on Cycle 1 Day 1
Description: The apparent terminal half-life was defined as the time required for the plasma concentration of drug to decrease 50% in the final stage of its elimination.
Time Frame: Cycle 1: Pre-morning dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8, hours post dose, pre-evening dose (Hour 12) at Day 1
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Arm/Group | Part 1: Pimasertib 30 mg in Solid Tumor | Part 1: Pimasertib 45 mg in Solid Tumor | Part 1: Pimasertib 60 mg in Solid Tumor | Part 1: Pimasertib 30 mg in HCC
Number analyzed (Participants) | 3 | 8 | 6 | 5
hours | 3.480 [3.43 to 4.78] | 3.545 [2.77 to 5.24] | 3.935 [2.71 to 5.61] | 4.560 [3.27 to 11.5]

18. Secondary Outcome: Apparent Terminal Half-life (t1/2) of Part 1: Pimasertib 45 mg in HCC Arm on Cycle 1 Day 1
Description: The apparent terminal half-life was defined as the time required for the plasma concentration of drug to decrease 50% in the final stage of its elimination. The summarized data was not available for this arm therefore individual data was presented.
Time Frame: Cycle 1: Pre-morning dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8, hours post dose, pre-evening dose (Hour 12) at Day 1
Population: as for outcome 4
Measure: Number; unit: hours
Arm/Group | Part 1: Pimasertib 45 mg in HCC
Number analyzed (Participants) | 2
hours
  Subject 1 | 5.68
  Subject 2 | 5.46

19. Secondary Outcome: Apparent Terminal Half-life (t1/2) of Pimasertib on Cycle 1 Day 15
Description: The apparent terminal half-life was defined as the time required for the plasma concentration of drug to decrease 50% in the final stage of its elimination. Data were not reported for "Part 1: Pimasertib 45 mg In HCC" arm as there were no PK samples collected for this arm.
Time Frame: Cycle 1: Pre-morning dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8, hours post dose, pre-evening dose (Hour 12) at Day 15
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Groups:
- Part 1: Pimasertib 30 mg in Solid Tumor: Subjects with solid tumor were administered with Pimasertib 30 mg BID until disease progression, intolerable toxicity, investigators decision to discontinue treatment or withdrawal of consent by the subject.
- Part 1: Pimasertib 45 mg in Solid Tumor: Subjects with solid tumor were administered with Pimasertib 45 mg BID until disease progression, intolerable toxicity, investigators decision to discontinue treatment or withdrawal of consent by the subject.
- Part 1: Pimasertib 60 mg in Solid Tumor: Subjects with solid tumor were administered with Pimasertib 60 mg BID until disease progression, intolerable toxicity, investigators decision to discontinue treatment or withdrawal of consent by the subject.
Arm/Group | Part 1: Pimasertib 30 mg in Solid Tumor | Part 1: Pimasertib 45 mg in Solid Tumor | Part 1: Pimasertib 60 mg in Solid Tumor | Part 1: Pimasertib 45 mg in HCC
Number analyzed (Participants) | 4 | 6 | 4 | 0
hours | 4.235 [0.775 to 5.21] | 4.000 [3.13 to 5.71] | 5.530 [2.92 to 8.24] |

20. Secondary Outcome: Apparent Terminal Half-life (t1/2) of Part 1: Pimasertib 30 mg in HCC Arm on Cycle 1 Day 15
Description: as for outcome 18
Time Frame: Cycle 1: Pre-morning dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8, hours post dose, pre-evening dose (Hour 12) at Day 15
Population: as for outcome 4
Measure: Number; unit: hours
Arm/Group | Part 1: Pimasertib 30 mg in HCC
Number analyzed (Participants) | 2
hours
  Subject 1 | 15.4
  Subject 2 | 5.41

21. Secondary Outcome: Apparent Clearance (CL/f) of Pimasertib on Cycle 1 Day 1
Description: Clearance of a drug was a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Apparent clearance after oral dose (CL/f) is influenced by the fraction absorbed.
Time Frame: Cycle 1: Pre-morning dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8, hours post dose, pre-evening dose (Hour 12) at Day 1
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter/hour (L/h)
Groups:
- Part 1: Pimasertib 60 mg in Solid Tumor: Subjects with HCC were administered with Pimasertib 60 mg BID in 21-day cycles until disease progression, intolerable toxicity, investigators decision to discontinue treatment or withdrawal of consent by the subject.
- Part 1: Pimasertib 30 mg in HCC: Subjects with HCC were administered with Pimasertib 30 mg BID until disease progression, intolerable toxicity, investigators decision to discontinue treatment or withdrawal of consent by the subject.
Arm/Group | Part 1: Pimasertib 30 mg in Solid Tumor | Part 1: Pimasertib 45 mg in Solid Tumor | Part 1: Pimasertib 60 mg in Solid Tumor | Part 1: Pimasertib 30 mg in HCC
Number analyzed (Participants) | 3 | 7 | 5 | 3
liter/hour (L/h) | 41.67 (80.5) | 48.17 (52.8) | 32.62 (54.6) | 32.19 (27.3)

22. Secondary Outcome: Apparent Clearance (CL/f) of Part 1: Pimasertib 45 mg in HCC Arm on Cycle 1 Day 1
Description: Clearance of a drug was a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Apparent clearance after oral dose (CL/f) is influenced by the fraction absorbed. The summarized data was not available for this arm therefore individual data was presented.
Time Frame: Cycle 1: Pre-morning dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8, hours post dose, pre-evening dose (Hour 12) at Day 1
Population: as for outcome 4
Measure: Number; unit: L/h
Arm/Group | Part 1: Pimasertib 45 mg in HCC
Number analyzed (Participants) | 2
L/h
  Subject 1 | 18.5
  Subject 2 | 23.7

23. Secondary Outcome: Apparent Clearance at Steady-state (CLss/f) of Pimasertib on Cycle 1 Day 15
Description: Apparent clearance at steady state was reported. Clearance of a drug was a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Data were not reported for "Part 1: Pimasertib 45 mg In HCC" arm as there were no PK samples collected for this arm.
Time Frame: Cycle 1: Pre-morning dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8, hours post dose, pre-evening dose (Hour 12) at Day 15
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Part 1: Pimasertib 30 mg in Solid Tumor | Part 1: Pimasertib 45 mg in Solid Tumor | Part 1: Pimasertib 60 mg in Solid Tumor | Part 1: Pimasertib 45 mg in HCC
Number analyzed (Participants) | 4 | 6 | 4 | 0
L/h | 25.24 (73.6) | 40.00 (62.1) | 28.02 (37.6) |

24. Secondary Outcome: Apparent Clearance at Steady-state (CLss/f) of Part 1: Pimasertib 30 mg in HCC Arm on Cycle 1 Day 15
Description: Apparent clearance at steady state was reported. Clearance of a drug was a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. The summarized data was not available for this arm therefore individual data was presented.
Time Frame: Cycle 1: Pre-morning dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8, hours post dose, pre-evening dose (Hour 12) at Day 15
Population: as for outcome 4
Measure: Number; unit: L/h
Arm/Group | Part 1: Pimasertib 30 mg in HCC
Number analyzed (Participants) | 2
L/h
  Subject 1 | 13.3
  Subject 2 | 17.8

25. Secondary Outcome: Apparent Volume of Distribution at Terminal Phase (Vz/f) of Pimasertib on Cycle 1 Day 1
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired serum concentration of a drug. Apparent volume of distribution after oral dose (Vz/f) was influenced by the fraction absorbed.
Time Frame: Cycle 1: Pre-morning dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8, hours post dose, pre-evening dose (Hour 12) at Day 1
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Part 1: Pimasertib 30 mg in Solid Tumor | Part 1: Pimasertib 45 mg in Solid Tumor | Part 1: Pimasertib 60 mg in Solid Tumor | Part 1: Pimasertib 30 mg in HCC
Number analyzed (Participants) | 3 | 7 | 5 | 3
liters | 231.2 (71.6) | 238.1 (46.7) | 169.8 (29.7) | 177.2 (15.9)

26. Secondary Outcome: Apparent Volume of Distribution at Terminal Phase (Vz/f) Part 1: Pimasertib 45 mg in HCC Arm on Cycle 1 Day 1
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired serum concentration of a drug. The summarized data was not available for this arm therefore individual data was presented.
Time Frame: Cycle 1: Pre-morning dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8, hours post dose, pre-evening dose (Hour 12) at Day 1
Population: as for outcome 4
Measure: Number; unit: liters
Arm/Group | Part 1: Pimasertib 45 mg in HCC
Number analyzed (Participants) | 2
liters
  Subject 1 | 152
  Subject 2 | 187

27. Secondary Outcome: Apparent Volume of Distribution at Terminal Phase (Vz/f) of Pimasertib on Cycle 1 Day 15
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired serum concentration of a drug. Apparent volume of distribution after oral dose (Vz/f) was influenced by the fraction absorbed. Data were not reported for "Part 1: Pimasertib 45 mg In HCC" arm as there were no PK samples collected for this arm.
Time Frame: Cycle 1: Pre-morning dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8, hours post dose, pre-evening dose (Hour 12) at Day 15
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Part 1: Pimasertib 30 mg in Solid Tumor | Part 1: Pimasertib 45 mg in Solid Tumor | Part 1: Pimasertib 60 mg in Solid Tumor | Part 1: Pimasertib 45 mg in HCC
Number analyzed (Participants) | 4 | 6 | 4 | 0
liters | 105.0 (161.1) | 233.9 (46.4) | 209.1 (10.6) |

28. Secondary Outcome: Apparent Volume of Distribution at Terminal Phase (Vz/f) of Part 1: Pimasertib 30 mg in HCC Arm on Cycle 1 Day 15
Description: as for outcome 26
Time Frame: Cycle 1: Pre-morning dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8, hours post dose, pre-evening dose (Hour 12) at Day 15
Population: as for outcome 4
Measure: Number; unit: liters
Arm/Group | Part 1: Pimasertib 30 mg in HCC
Number analyzed (Participants) | 2
liters
  Subject 1 | 297
  Subject 2 | 139

29. Secondary Outcome: Accumulation Ratio for AUC Racc(AUC) of Pimasertib
Description: Racc (AUC) was calculated as, area under the curve from time zero to end of dosing interval on Day 1 divided by area under the curve from time zero to end of dosing interval on Day 15. Data were not reported for "Part 1: Pimasertib 45 mg In HCC" arm as there were no PK samples collected for this arm.
Time Frame: Cycle 1: Pre-morning dose, 0.5, 1, 1.5, 2, 2.5, 4, 6, 8, hours post dose, pre-evening dose (Hour 12) at Day 1 and Day 15
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Part 1: Pimasertib 30 mg in Solid Tumor | Part 1: Pimasertib 45 mg in Solid Tumor | Part 1: Pimasertib 60 mg in Solid Tumor | Part 1: Pimasertib 45 mg in HCC
Number analyzed (Participants) | 3 | 6 | 4 | 0
ratio | 1.782 (4.2) | 1.382 (30.2) | 1.311 (51.5) |

30. Secondary Outcome: Accumulation Ratio for AUC Racc(AUC) of Part 1: Pimasertib 30 mg In HCC Arm
Description: Racc (AUC) was calculated as, area under the curve from time zero to end of dosing interval on Day 1 divided by area under the curve from time zero to end of dosing interval on Day 15.
Time Frame: as for outcome 29
Population: as for outcome 4
Measure: Number; unit: ratio
Arm/Group | Part 1: Pimasertib 30 mg in HCC
Number analyzed (Participants) | 2
ratio
  Subject 1 | 2.43
  Subject 2 | 1.83

31. Secondary Outcome: Accumulation Ratio for Cmax Racc(Cmax) of Pimasertib
Description: Racc (Cmax) was calculated as, maximum observed plasma concentration on Day 1 (Cmax) divided by maximum observed plasma concentration on Day 15 (Cmax). Data were not reported for "Part 1: Pimasertib 45 mg In HCC" arm as there were no PK samples collected for this arm.
Time Frame: as for outcome 29
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Part 1: Pimasertib 30 mg in Solid Tumor | Part 1: Pimasertib 45 mg in Solid Tumor | Part 1: Pimasertib 60 mg in Solid Tumor | Part 1: Pimasertib 45 mg in HCC
Number analyzed (Participants) | 4 | 6 | 5 | 0
ratio | 1.227 (38.3) | 0.8281 (65.5) | 1.215 (61.3) |

32. Secondary Outcome: Accumulation Ratio for Cmax Racc(Cmax) of Part 1: Pimasertib 30 mg In HCC Arm
Description: Racc (Cmax) was calculated as, maximum observed plasma concentration on Day 1 (Cmax) divided by maximum observed plasma concentration on Day 15 (Cmax).
Time Frame: as for outcome 29
Population: as for outcome 4
Measure: Number; unit: ratio
Arm/Group | Part 1: Pimasertib 30 mg in HCC
Number analyzed (Participants) | 2
ratio
  Subject 1 | 1.50
  Subject 2 | 2.31

33. Secondary Outcome: Percentage of Subjects With Best Overall Response
Description: Percentage of subjects with best overall response in each category (complete response [CR], partial response [PR], stable disease [SD], progressive disease [PD]) according to Response Evaluation Criteria in Solid Tumors (RECIST Version 1.1) was reported. CR was defined as disappearance of all target and all non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study) or unequivocal progression of existing non-target lesions. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Day 1 of Cycle 3 and Day 1 of every alternate until end of treatment (up to a maximum of 35.4 weeks)
Population: Efficacy analysis set included all subjects who received at least one administration of planned dose of pimasertib and who have had at least one efficacy assessment after the first dose.
Measure: Number; unit: percentage of subjects
Groups:
- Part 1: Pimasertib 45 mg in HCC: Subjects with HCC were administered with Pimasertib 45 mg BID until disease progression, intolerable toxicity, investigators decision to discontinue treatment or withdrawal of consent by the subject.
Arm/Group | Part 1: Pimasertib 30 mg in Solid Tumor | Part 1: Pimasertib 45 mg in Solid Tumor | Part 1: Pimasertib 60 mg in Solid Tumor | Part 1: Pimasertib 30 mg in HCC | Part 1: Pimasertib 45 mg in HCC
Number analyzed (Participants) | 3 | 7 | 4 | 4 | 2
percentage of subjects
  CR | 0 | 0 | 0 | 0 | 0
  PR | 0 | 42.9 | 0 | 0 | 0
  SD | 0 | 14.3 | 0 | 0 | 0
  PD | 66.7 | 42.9 | 75.0 | 75.0 | 50.0
  Not evaluable | 33.3 | 0 | 25.0 | 25.0 | 50.0

34. Secondary Outcome: Percentage of Subjects With Objective Response
Description: Percentage of subjects with objective response (CR plus PR) according to RECIST Version 1.1 was reported. CR was defined as disappearance of all target and all non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Day 1 of Cycle 3 and Day 1 of every alternate until end of treatment (up to a maximum of 35.4 weeks)
Population: Efficacy analysis set' included all subjects who received at least one administration of planned dose of pimasertib and who have had at least one efficacy assessment after the first dose.
Measure: Number; unit: percentage of subjects
Groups:
- Part 1: Pimasertib 30 mg in Solid Tumor: Subjects with solid tumor were administered with Pimasertib 30 mg twice a day (BID) until disease progression, intolerable toxicity, investigators decision to discontinue treatment or withdrawal of consent by the subject.
- Part 1: Pimasertib 30 mg in HCC; Part 1: Pimasertib 45 mg in HCC: Subjects with HCC were administered with Pimasertib 45 mg BID until disease progression, intolerable toxicity, investigators decision to discontinue treatment or withdrawal of consent by the subject.
Arm/Group | Part 1: Pimasertib 30 mg in Solid Tumor | Part 1: Pimasertib 45 mg in Solid Tumor | Part 1: Pimasertib 60 mg in Solid Tumor | Part 1: Pimasertib 30 mg in HCC | Part 1: Pimasertib 45 mg in HCC
Number analyzed (Participants) | 3 | 7 | 4 | 4 | 2
percentage of subjects | 0 | 42.9 | 0 | 0 | 0

35. Secondary Outcome: Percentage of Subjects With Disease Control
Description: Percentage of subjects with disease control (CR plus PR plus greater than 12 weeks SD) according to RECIST Version 1.1 was reported CR was defined as disappearance of all target and all non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study) or unequivocal progression of existing non-target lesions.
Time Frame: Day 1 of Cycle 3 and Day 1 of every alternate until end of treatment (up to a maximum of 35.4 weeks)
Population: as for outcome 33
Measure: Number; unit: percentage of subjects
Arm/Group | Part 1: Pimasertib 30 mg in Solid Tumor | Part 1: Pimasertib 45 mg in Solid Tumor | Part 1: Pimasertib 60 mg in Solid Tumor | Part 1: Pimasertib 30 mg in HCC | Part 1: Pimasertib 45 mg in HCC
Number analyzed (Participants) | 3 | 7 | 4 | 4 | 2
percentage of subjects | 0 | 57.1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 30 days post last dose of study drug; assessed maximum up to 39.4 weeks
Arm/Group | Part 1: Pimasertib 30 mg in Solid Tumor | Part 1: Pimasertib 45 mg in Solid Tumor | Part 1: Pimasertib 60 mg in Solid Tumor | Part 1: Pimasertib 30 mg in HCC | Part 1: Pimasertib 45 mg in HCC
Serious Adverse Events (participants affected / at risk) | 2/4 | 2/9 | 2/6 | 2/5 | 0/2
Other Adverse Events (participants affected / at risk) | 4/4 | 9/9 | 6/6 | 5/5 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Pimasertib 30 mg in Solid Tumor (N=4) | Part 1: Pimasertib 45 mg in Solid Tumor (N=9) | Part 1: Pimasertib 60 mg in Solid Tumor (N=6) | Part 1: Pimasertib 30 mg in HCC (N=5) | Part 1: Pimasertib 45 mg in HCC (N=2)
Disease progression (General disorders) | 1 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 2 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Liver disorder (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Pimasertib 30 mg in Solid Tumor (N=4) | Part 1: Pimasertib 45 mg in Solid Tumor (N=9) | Part 1: Pimasertib 60 mg in Solid Tumor (N=6) | Part 1: Pimasertib 30 mg in HCC (N=5) | Part 1: Pimasertib 45 mg in HCC (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Pericardia effusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Retinal detachment (Eye disorders) | 3 | 6 | 5 | 3 | 1
Vision blurred (Eye disorders) | 3 | 6 | 5 | 3 | 1
Retinal haemorrhage (Eye disorders) | 0 | 2 | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 1 | 1 | 0 | 0
Macular oedema (Eye disorders) | 0 | 0 | 1 | 1 | 0
Ocular hypertension (Eye disorders) | 0 | 1 | 0 | 0 | 0
Retinal tear (Eye disorders) | 0 | 1 | 0 | 0 | 0
Macular detachment (Eye disorders) | 0 | 0 | 0 | 1 | 0
Metamorphopsia (Eye disorders) | 0 | 0 | 0 | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 1 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 5 | 3 | 3 | 1
Nausea (Gastrointestinal disorders) | 1 | 3 | 2 | 2 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 4 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 3 | 1 | 2
Constipation (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 1 | 5 | 4 | 0 | 1
Pyrexia (General disorders) | 1 | 2 | 3 | 2 | 0
Localised oedema (General disorders) | 0 | 2 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 2 | 1 | 1
Malaise (General disorders) | 1 | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 1 | 1
Feeling hot (General disorders) | 0 | 0 | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Contrast media allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Frostbite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 4 | 6 | 5 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 5 | 1 | 2 | 1
Alanine aminotransferase increased (Investigations) | 2 | 2 | 1 | 2 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 1 | 1 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 2 | 0 | 1 | 0
Blood creatine phosphokinase MB increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0 | 0 | 0
Fibrin D dimer increased (Investigations) | 0 | 1 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 2 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 4 | 3 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 2 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 6 | 3 | 4 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 3 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 2 | 1 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Due to the Sponsor's decision not to pursue the study drug as monotherapy, the Expansion Phase (Part 2) of the study was not conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No